CLINICAL TRIAL: NCT03676608
Title: Study of Health Education to Improve Adherence to Breastfeeding in Primiparous Women Through the Use of Bee Wax Mammary Areolae
Brief Title: Use of Bee Wax Mammary Areolae to Improve Breastfeeding
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alicante (Other)
Responsible Party: Principal Investigator, María Mercedes Rizo-Baeza, Professor, University of Alicante
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UA-2014-11-12
Record Dates: First submitted 2018-06-29; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bee wax mammary areolae (Experimental): Usual educational care plus the product.
  The product to be valued are mammary areolae made by hand with organic beeswax. Despite its honey aroma, it does not contain honey. The wax used for the manufacture of the areolae is operculum. This wax is used and not another because it avoids possible residues and allergies that may contain other types of waxes. The operculum wax is used as a thickener in pharmacy and cosmetic products as a fat base in ointments and creams.
  Interventions: Biological: Bee Wax Mammary Areolae; Other: Usual educational care
- Control (Active Comparator): Usual educational care.
  Interventions: Other: Usual educational care

INTERVENTIONS:
Biological: Bee Wax Mammary Areolae — The product to be valued are mammary areolae made by hand with organic beeswax. Despite its honey aroma, it does not contain honey. The wax used for the manufacture of the areolae is operculum. This wax is used and not another because it avoids possible residues and allergies that may contain other types of waxes. The operculum wax is used as a thickener in pharmacy and cosmetic products as a fat base in ointments and creams.
  Arms: Bee wax mammary areolae
Other: Usual educational care — The WHO protocol for maternal lactation.

SUMMARY:
A comparative randomized intervention study is presented between a mixed strategy of use of bee wax mammary areolae. Together with the health education program for the promotion of breastfeeding by the WHO and another educational program with the aim of improving the adherence of breastfeeding to primiparous women. The use of both interventions can contribute to the adherence to exclusive maternity in 20% in the first 6 months of life, than only with the educational program.

The study provides evidence of nursing practice, thus contributing to the improvement of nursing mothers in the prevention of lesions in the nipple and care in them if they occur. Consequently, improve the rates of successful breastfeeding, as well as the quality of life of breastfeeding mothers. The study will be carried out with several groups of midwives in Health Centers, in Spain, Colombia and Mexico. The sample was calculated in 240 women who attend the midwife's controls between week 29 and 40.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women regardless of age.
* Attended in the consultation of midwives of health centers selected for the study.
* Signature of informed consent.

Exclusion Criteria:

* Atopias and dermatological problems.
* No willingness to continue breastfeeding.
* Mental diseases.
* Allergy to the products of the bee.
* No informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Primiparaous women.
Enrollment: 240 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of women with exclusive breastfeeding for 6 months. | 6 months
Exclusive breastfeeding time in days. | 6 months

SECONDARY OUTCOMES:
Mammary congestion | 6 months
  This is measured by the clinical diagnosis.
Mastitis | 6 months
  This is measured by the clinical diagnosis.
Cracks | 6 months
  This is measured by the clinical diagnosis.
Irritation | 6 months
  This is measured by the clinical diagnosis.

CONTACTS AND LOCATIONS:
Locations (3):
- Universidad Simón Bolívar, Barranquilla, Colombia
- Universidad Autónoma de Nuevo León, San Nicolás de los Garza, Nuevo León, Mexico
- University of Alicante, San Vicent del Raspeig, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
The data will not be publicly available.

REFERENCES:
- [Background] Vieira F, Bachion MM, Mota DD, Munari DB. A systematic review of the interventions for nipple trauma in breastfeeding mothers. J Nurs Scholarsh. 2013 Jun;45(2):116-25. doi: 10.1111/jnu.12010. Epub 2013 Mar 1. PMID 23452043
- [Background] Britton C, McCormick FM, Renfrew MJ, Wade A, King SE. Support for breastfeeding mothers. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD001141. doi: 10.1002/14651858.CD001141.pub3. PMID 17253455